CLINICAL TRIAL: NCT01101711
Title: Endocrine Dysfunction and Quality of Life After Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Erik Kronvall, Dr., Lund University Hospital
Other Study IDs: 65/2006
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Endocrine Dysfunction; Cerebral Infarctions; Quality of Life
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with subarachnoid hemorrhage

SUMMARY:
Investigation of the incidence of endocrine dysfunction following subarachnoid hemorrhage (SAH), and to see if this has a relation to CNS lesions as evaluated by MRI and to common symptoms after SAH such as general exhaustion, lack of initiative, increased sleep demand and reduced quality of life.

ELIGIBILITY:
Inclusion Criteria:

* acute aneurysmal subarachnoid hemorrhage

Exclusion Criteria:

* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the southern part of Sweden who have suffered subarachnoid hemorrhage and admitted to the Department of Neurosurgery in Lund
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-11; Primary Completion 2011-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Lund, Sweden